CLINICAL TRIAL: NCT00700999
Title: Neurofunctional Markers of SSRI Treatment Response in PTSD
Brief Title: Brain Markers of Treatment Response in Post-Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MHBA-002-08S
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Other): Intervention-Paroxetine
  Interventions: Drug: Paroxetine
- Arm 2 (No Intervention): No Intervention

INTERVENTIONS:
Drug: Paroxetine — Paroxetine 20-40mg po QD for 12 weeks
  Other Names: Paxil (brand name)
  Arms: Arm 1

SUMMARY:
The purpose of this study is to examine if treatment of post-traumatic stress disorder in combat veterans with paroxetine changes brain responses as measured by functional magnetic resonance imaging and if brain responses can predict who will get better with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with clinical diagnosis of post-traumatic stress disorder from combat related to deployment to Afghanistan/Iraq (Operation Enduring Freedom/Operation Iraqi Freedom)

Exclusion Criteria:

* Intolerance or sensitivity to paroxetine
* Major medical or neurologic illness
* Current psychotropic medication or active psychotherapy treatment
* Other major psychiatric illness

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2008-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K. Luan Phan, MD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (3):
- United States (3):
  - Jesse Brown VA Medical Center Community-Based Outpatient Clinic Lake Side Divison, Chicago, IL, Chicago, Illinois
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in this study from 3/1/09 to 12/31/11. Participants were recruited by flyers in the community and within the Ann Arbor Veterans Affairs Health System and through professional referrals within the Ann Arbor Veterans Affairs Health System through the outpatient psychiatry clinics and primary care clinics.
Pre-assignment Details: All participants went through an initial screening visit in which they signed the informed consent document and completed multiple assessments and a medical evaluation in order to assure that they were able to participate in the study and that they did not meet any exclusionary conditions.
Groups:
- Treatment (Paroxetine) Group: Veterans returning from OEF/OIF with documented exposure to combat trauma who meet criteria for DSM-IV diagnosis of PTSD. Completed 12 weeks of treatment with paroxetine (20-40mg QD)
- Combat Exposed Controls: Veterans returning from OEF/OIF with documented exposure to combat trauma who do not meet criteria for DSM-IV diagnosis of PTSD
Period: Overall Study
Arm/Group | Treatment (Paroxetine) Group | Combat Exposed Controls
Started | 36 | 29
First MRI Scan | 29 | 22
Second MRI Scan | 19 | 18
Completed | 21 | 20
Not Completed | 15 | 9
Not completed — Lost to Follow-up | 7 | 7
Not completed — Excluded - did not meet study criteria | 0 | 1
Not completed — Withdrawal by Subject | 8 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Participants have been determined by the number of participants that completed the first MRI scan.
Groups:
- Treatment Group: Veterans returning from OEF/OIF with documented exposure to combat trauma who meet criteria for DSM-IV diagnosis of PTSD
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Combat Exposed Controls | Total
Number analyzed (Participants) | 29 | 22 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 22 | 51
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 29 | 21 | 50
Region of Enrollment [Number; unit: participants]
  United States | 29 | 22 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Brain Response Measured by Functional Magnetic Resonance Imaging (fMRI)
Description: Mean percent change in brain response in the prefrontal cortex during an emotion reappraisal task in the treatment (paroxetine) group and in the Combat Exposed Control group. Target areas are analyzed from fMRI scans which were completed before participants receive treatment and again after participants received 12 weeks of treatment with paroxetine (20-40mg QD). Combat Exposed Control participants received an fMRI scan after signing initial consent and again 12 weeks later.
Time Frame: Baseline and 12 weeks
Population: The number of participants analyzed is only 17 in each arm. The total number of participants in the Intervention group who completed fMRI scans pre-treatment and post treatment is only 19, in the Combat Exposed Control Group it is 18. Three of the participants scans were removed from data analysis due to the level of movement during the scan.
Measure: Mean (Standard Deviation); unit: percent change in BOLD signal
Groups:
- Treatment (Paroxetine) Group: Veterans returning from OEF/OIF with documented exposure to combat trauma who meet criteria for DSM-IV diagnosis of PTSD
- Combat Exposed Control: Veterans returning from OEF/OIF with documented exposure to combat trauma who do not meet criteria for DSM-IV diagnosis of PTSD.
Arm/Group | Treatment (Paroxetine) Group | Combat Exposed Control
Number analyzed (Participants) | 17 | 17
percent change in BOLD signal | -.92 (0.90) | .07 (1.78)
Statistical Analysis 1: Comparison: Treatment (Paroxetine) Group; Test type: Superiority or Other; p = .001, t-test, 2 sided; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-1.38 to -0.45], Standard Deviation 0.90
Statistical Analysis 2: Comparison: Combat Exposed Control; Test type: Superiority or Other; p = .869, t-test, 2 sided; Mean Difference (Final Values) = .07, 95% CI 2-sided [-.84 to .99], Standard Deviation 1.78

ADVERSE EVENTS:
Description: In the adverse events described below the total number of participants at risk for other adverse events is not consistent with the total number of participants at risk for other adverse events in the Arms/Groups i.e., "36" and "29" respectively. The numbers are correct due to only 22 participants having participated in the fMRI scans.
Arm/Group | Treatment (Paroxetine) Group | Combat Exposed Controls
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/29
Other Adverse Events (participants affected / at risk) | 28/36 | 1/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment (Paroxetine) Group (N=36) | Combat Exposed Controls (N=29)
Psychological/Emotional Adverse Event (Psychiatric disorders) | 5/28 (5) | 0 (0) — Increased anxiety reported at the study visit. Empathic listening, supportive responding provided. Unclear if increase in anxiety symptoms related to PTSD illness, current psychosocial stressors, and/or medication. No specific terms were collected.
Anxiety experience during fMRI scanning (Psychiatric disorders) | 2/29 (2) | 1/22 (1) — Increased anxiety per subject report; Empathic listening & supportive responding was provided. The subject's mood & psychological/psychiatric symptoms did not warrant "ongoing psychotherapy treatment of any kind" beyond what was offered in the study
Physical Side Effect to Medication - Blurred Vision (Psychiatric disorders) | 8 (8) | 0/0 (0)
Physical Side Effect to Medication - Chest Pain (Psychiatric disorders) | 7 (7) | 0/0 (0)
Physical Side Effect to Medication - Constipation (Psychiatric disorders) | 8 (8) | 0/0 (0)
Physical Side Effect to Medication - Diarrhea (Psychiatric disorders) | 9 (9) | 0/0 (0)
Physical Side Effect to Medication - Difficulty Urinating (Psychiatric disorders) | 2 (2) | 0/0 (0)
Physical Side Effect to Medication - Difficulty with erections or sexual functioning (Psychiatric disorders) | 17 (17) | 0/0 (0)
Physical Side Effect to Medication - Dizziness (Psychiatric disorders) | 13 (13) | 0/0 (0)
Physical Side Effect to Medication - Drowsiness (Psychiatric disorders) | 24 (24) | 0/0 (0)
Physical Side Effect to Medication - Dry mouth (Psychiatric disorders) | 14 (14) | 0/0 (0)
Physical Side Effect to Medication - Feeling that familiar things are strange or unreal (Psychiatric disorders) | 9 (9) | 0/0 (0)
Physical Side Effect to Medication - Headaches (Psychiatric disorders) | 24 (24) | 0/0 (0)
Physical Side Effect to Medication - Heart pounding or racing (Psychiatric disorders) | 20 (20) | 0/0 (0)
Physical Side Effect to Medication - Hot or cold spells (Psychiatric disorders) | 11 (11) | 0/0 (0)
Physical Side Effect to Medication - Increased salivation (Psychiatric disorders) | 2 (2) | 0/0 (0)
Physical Side Effect to Medication - Nausea (Psychiatric disorders) | 17 (17) | 0/0 (0)
Physical Side Effect to Medication - Nervousness (Psychiatric disorders) | 18 (18) | 0/0 (0)
Physical Side Effect to Medication - Numbness or tingling (Psychiatric disorders) | 15 (15) | 0/0 (0)
Physical Side Effect to Medication - Overeating (Psychiatric disorders) | 12 (12) | 0/0 (0)
Physical Side Effect to Medication - Panic (Psychiatric disorders) | 13 (13) | 0/0 (0)
Physical Side Effect to Medication - Poor Appetite (Psychiatric disorders) | 17 (17) | 0/0 (0)
Physical Side Effect to Medication - Soreness (Psychiatric disorders) | 23 (23) | 0/0 (0)
Physical Side Effect to Medication - Sweating (Psychiatric disorders) | 15 (15) | 0/0 (0)
Physical Side Effect to Medication - Tense (Psychiatric disorders) | 25 (25) | 0/0 (0)
Physical Side Effect to Medication - Trembling (Psychiatric disorders) | 12 (12) | 0/0 (0)
Physical Side Effect to Medication - Trouble falling asleep (Psychiatric disorders) | 25 (25) | 0/0 (0)
Physical Side Effect to Medication - Trouble getting your breath (Psychiatric disorders) | 8 (8) | 0/0 (0)
Physical Side Effect to Medication - Trouble remembering things (Psychiatric disorders) | 26 (26) | 0/0 (0)
Physical Side Effect to Medication - Trouble staying asleep (Psychiatric disorders) | 24 (24) | 0/0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes